CLINICAL TRIAL: NCT06898177
Title: Development and Testing of a Mobile App to Scale Delivery of Cognitive-behavioral Therapy for Avoidant/Restrictive Food Intake Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Paraskevi E. Kambanis, Clinical Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025P000075
Record Dates: First submitted 2025-03-18; First posted 2025-03-27 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Avoidant/Restrictive Food Intake Disorder (ARFID)
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mCBT-AR (Experimental)
  Interventions: Behavioral: mCBT-AR
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: mCBT-AR — mCBT-AR is an 8-week virtual treatment for avoidant/restrictive food intake disorder delivered via mobile application
  Arms: mCBT-AR

SUMMARY:
Avoidant/restrictive food intake disorder (ARFID) is a serious and impairing eating disorder - occurring in up to 4% of adults - for which most individuals do not have access to treatment. The proposed study aims to develop and test a mobile app to scale delivery of cognitive-behavioral therapy for ARFID. Knowledge gained will contribute to the development of a clinically accessible, scalable, inexpensive treatment for ARFID, a highly impairing disorder for which there are significant barriers to care access.

ELIGIBILITY:
Inclusion Criteria:

1. Current avoidant/restrictive food intake disorder based on DSM-5 criteria
2. Must not have completed face-to-face CBT-AR at the Eating Disorders Clinical and Research Program at Massachusetts General Hospital
3. Ability to speak, write, and understand English
4. Residence in the United States
5. Access to an internet-connected smartphone device

Exclusion Criteria:

1. Underweight status (i.e., BMI < 18.5 kg/m2)
2. Complete lack of oral intake or dependence on supplemental feeding
3. Feeding or eating disorder other than ARFID
4. Any comorbid clinically significant disorder that would require attention beyond the study treatment

6. Medical instability requiring inpatient care according to the American Psychiatric Association 2023 treatment guidelines for eating disorders 7. Medical history of intellectual disability 8. Illiteracy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2030-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Pica, ARFID, and Rumination Disorder Interview - ARFID Questionnaire (PARDI-AR-Q) | Change from baseline (assessed at study entry) to final session, which occurs an average of eight weeks after baseline (measured at weekly study treatment sessions)
  The PARDI-AR-Q is a 32-item self-report measure based on the Pica, ARFID, and Rumination Disorder Interview that assesses ARFID diagnostic criteria and the presence and severity of each ARFID profile. Severity scores for each profile range from 0-6, with higher scores indicating greater severity.
Food Neophobia Scale (FNS) | Change from baseline (assessed at study entry) to final session, which occurs an average of eight weeks after baseline (measured at weekly study treatment sessions)
  The Food Neophobia Scale is a 6-item measure that measures reluctance to try new foods. Scores range from 7-42. Higher scores on the FNS are indicative of greater behavioral responses to novel foods.